CLINICAL TRIAL: NCT05330390
Title: Study on the Population Pharmacokinetics and Individualized Administration of Levetiracetam in Epileptic Patients With Diabetic Kidney Disease
Brief Title: Study on the Population Pharmacokinetics of Levetiracetam in Epileptic Patients With Diabetic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: byssc1985-2022
Record Dates: First submitted 2022-04-03; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy; Diabetic Nephropathy
Keywords: Levetiracetam; Population pharmacokinetics
MeSH Terms: conditions — Epilepsy; Diabetic Nephropathies | interventions — Levetiracetam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Levetiracetam — Epilepsy, treatment with levetiracetam

SUMMARY:
The individualized drug delivery system of levetiracetam based on population pharmacokinetics and quantitative pharmacology model in patients with epilepsy complicated by diabetic kidney disease was established. To clarify the clinical feasibility of model-based individualized drug administration scheme.

DETAILED DESCRIPTION:
A quantitative pharmacological model for the development of levetiracetam in epileptic patients with diabetic nephropathy is proposed. First, a model based active levetiracetam based individualized initial dose regimen was established by using clinical simulation techniques. A simulation model was established for patients with diabetes mellitus and kidney disease, including information on patients' gender, age and other factors, diabetes mellitus, renal disease history, creatinine clearance rate, glomerular filtration rate, urinary protein level and blood lipid level. Secondly, the simulated clinical trial combining simulation model and population pharmacokinetic model is used to compare the compliance rate of levetiracetam blood concentration in patients with different dose treatment schemes, so as to obtain the optimal individualized administration scheme. Finally, Bayesian feedback technology is used to improve the passive dose adjustment scheme, and model-based Bayesian feedback technology is used to establish a dose adjustment scheme based on area under curve (AUC), so as to clarify the optimal blood sampling scheme and monitoring method.

ELIGIBILITY:
Inclusion Criteria:

- Patients with seizures and diabetic nephropathy who were treated with levetiracetam.

Exclusion Criteria:

* patients who rejected

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The method of continuous and non random enrollment was adopted.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-04 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood drug concentration | through study completion, an average of 1 year
  After treating with levetiracetam, blood samples were collected at different time periods

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shandong University, Jinan, Shandong, China